CLINICAL TRIAL: NCT03720080
Title: Observational Study to Compare Adaptions of Basal Rate Doses Using Self-build OpenAPS Artificial Pancreas Compared With Medtronic 670G Hybrid Closed Loop in Type 1 Diabetes
Brief Title: The OpenAPS_ShadowMode Study
Status: Terminated | Type: Observational
Why Stopped: Enough information was gathered in order to answer the primary research question
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: CUI_003
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Type1diabetes
Keywords: Type 1 Diabetes; Artificial Pancreas; Medtronic 670G; OpenAPS
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 670G/OpenAPS: Participants with Type 1 Diabetes wearing a Medtornic Minimed 670G hybrid closed loop system in parallel with a non-insulin injecting, self-constructed OpenAPS system.
  Interventions: Device: OpenAPS

INTERVENTIONS:
Device: OpenAPS — A self-constructed OpenAPS system will be worn contemporaneously to a Medtronic Minimed 670G hybrid closed loop system. Both systems will calculate recommended basal rate insulin adjustments but only the Minimed 670G system will inject insulin. The maximum treatment period will be 2 weeks per patient

SUMMARY:
The "Open Artificial Pancreas System (OpenAPS)" was designed to quickly spread technology and knowledge about the construction of artificial pancreas systems to patients with diabetes without awaiting clinical regulatory approval. OpenAPS is based on a privately shared software programs and available insulin pumps and glucose sensors. OpenAPS includes a "decision making" algorithm, which issues adaptions of basal rates to insulin pumps, which represents all fundamental aspects of closed loop artificial pancreas systems. The present study aims to compare the accuracy and performance of a self-constructed OpenAPS system with the approved hybrid closed loop system Medtronic Minimed 670G.

While wearing the Medtronic Minimed 670G in automode, study participants will wear an OpenAPS system in parallel, which does calculate basal rate adaptions based on continuous glucose monitoring data and its respective algorithm. The investigators aim to recruit 15 participants in an open label, single-center, single-arm, observational study. Insulin injection will only be provided by the Medtronic 670G HCL system (Basal rate insulin). The OpenAPS system will be worn contemporaneously, calculate recommended basal rate insulin adjustments but will not inject insulin. The maximum treatment period will be 2 weeks per patient.

DETAILED DESCRIPTION:
Insulin titration remains a demanding challenge in the treatment of type 1 diabetes mellitus (T1DM). The two most significant advances in terms of insulin dosing where the introduction of continuous subcutaneous insulin infusion (CSII) and continuous glucose monitoring (CGM) sensors. CSII allows to diligently titrate hourly basal rates of insulin, which tremendously increased insulin and meal-time flexibility. CGM sensors provide continuous documentation of glycemic excursions without the need for patients' activity.

The most recent development was to enable communication and data sharing between CSII and CGMS. The idea was to create an autonomous system that measured current glucose concentrations and issued an adequate insulin dose to the CSII device. These systems were entitled "closed loop systems" or "artificial pancreas" (AP).

In general, APs have three components: the CSII device, a CGM sensor, and a "decision-making" algorithm integrated in a microprocessor.

In 2006, the Juvenile Diabetes Research Foundation (JDRF) launched the "AP Project" and has been funding development in this area since that time. In 2013, the threshold suspend feature was approved by the American Food and Drug Administration (FDA) as part of the MiniMed 530G CSII and Enlite sensor CGM. Threshold suspend autonomously stopped basal rate insulin infusion if hypoglycaemia was imminent. It is categorized as hybrid closed loop (HCL) AP system. HCL autonomous adjusts basal rate insulin infusion yet requires active bolus application by the patient. Several trials confirmed its safety and efficacy in children and adults with type 1 diabetes. In clinical trials, general safety was high, glycemic control increased and the incidence of hypoglycaemia was significantly reduced. Based on these promising data, the FDA approved the Medtronic 670G as the first HCL automated insulin delivery system in the United States. In 2018, Medtronic 670G was approved in the European Union and in Switzerland for the treatment of patients with T1DM.

In 2013, an initiative called the "Open Artificial Pancreas System (OpenAPS)" gained significant attention in the diabetes community.(9) OpenAPS was designed to quickly spread AP technology to patients with diabetes without awaiting clinical trials and FDA approval. OpenAPS is based on a privately shared software program, which enables access and transfer of CGM data to a data cloud, the so called "Nightscout" software. Soon thereafter, the "Do-It-Yourself Pancreas System" (DIYPS) software was created. DIYPS is a "decision making" algorithm for insulin delivery. DIYPS was combined with the Nightscout-software and allowed communication between Medtronic CSII and CGM sensors, data retrieval and issuance of insulin-dosing. With this update, the DIYPS system and Nightscout-software together became a hybrid closed loop AP system, better known as "OpenAPS".

In Switzerland, OpenAPS gained considerable interest in technique-affine patients with T1DM, and there already are patients with T1DM using openAPS at our department, despite the recommendation to use only approved medical devices. The number of patients using OpenAPS might be small at the moment but is growing, and diabetes care experts are asked to respond to this trend. It is necessary to evaluate safety of OpenAPS in diabetes, which are free of charge, to be used "at your own risk", but regulate sensible parameters like insulin dosing in the treatment of diabetes.

The aim of the present study is to evaluate accuracy and performance of an individually build OpenAPS in the fasting and the postprandial state and to compare each step of dose titration with the Medtronic 670G system as an approved HCL reference system.

The investigators aim to recruit 15 participants in an open label, single-center, single-arm, observational study. Insulin injection will only be provided by the Medtronic 670G HCL system (Basal rate insulin). The OpenAPS system will be worn contemporaneously, calculate recommended basal rate insulin adjustments but will not inject insulin. The maximum treatment period will be 2 weeks per patient.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Aged ≥ 18 years
* T1D as defined by WHO for at least 1 year
* Planned use of the Medtronic 670G HCL system

Exclusion Criteria:

* Type 2 diabetes mellitus
* Gestational diabetes mellitus
* Participation in another trial which may in the opinion of the investigator interfere with the software algorithm
* Any mental condition rendering the patient incapable of giving informed consent
* Any disease or condition which in the opinion of the investigator would interfere with the trial performance and/or the physical and/or psychosocial safety of the study participant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with Type 1 Diabetes of both sexes, aged 18 to 75 years, who are treated in our Diabetes outpatient clinics and who are intented to use the Medtronic Minimed 670G hybrid closed loop system.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Adjustments of basal rate insulin infusion OpenAPS | Maximum duration of 2 weeks per participant
  Dose adjustments of basal rate insulin infusion calculated by OpenAPS during the study period
Adjustments of basal rate insulin infusion 670G | Maximum duration of 2 weeks per participant
  Dose adjustments of basal rate insulin infusion calculated by Minimed 670G during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Stettler, Prof MD, Study Director — Inselspital, Bern University Hospital, University of Bern
Locations (1):
- Universitätspoliklinik für Endokrinologie, Diabetologie und Klinische Ernährung, Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lewis D. Setting Expectations for Successful Artificial Pancreas/Hybrid Closed Loop/Automated Insulin Delivery Adoption. J Diabetes Sci Technol. 2018 Mar;12(2):533-534. doi: 10.1177/1932296817730083. Epub 2017 Sep 18. No abstract available. PMID 28918653
- [Background] Litchman ML, Lewis D, Kelly LA, Gee PM. Twitter Analysis of #OpenAPS DIY Artificial Pancreas Technology Use Suggests Improved A1C and Quality of Life. J Diabetes Sci Technol. 2019 Mar;13(2):164-170. doi: 10.1177/1932296818795705. Epub 2018 Sep 10. PMID 30198751
- [Result] Lewis D, Leibrand S; #OpenAPS Community. Real-World Use of Open Source Artificial Pancreas Systems. J Diabetes Sci Technol. 2016 Nov 1;10(6):1411. doi: 10.1177/1932296816665635. Print 2016 Nov. No abstract available. PMID 27510442
- See also: Official Website of the OpenAPS developer and community — https://openaps.org/